CLINICAL TRIAL: NCT01778478
Title: Pilot Study to Extend the K-SADS-PL to Adolescents and Young Adults
Brief Title: A Pilot Study to Extend the K-SADS-PL to Adolescents and Young Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130019; 13-M-0019
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-05-23

CONDITIONS: Depression; Anxiety Disorder; Cancer
Keywords: Anxiety; Depression; Adolescents and Adults; Cancer Diagnosis
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- An interview called the Schedule for Affective Disorders and Schizophrenia for School Age Children Present and Lifetime version (K-SADS-PL) is used to identify mental health problems among children and younger teens. Both the child and a parent are asked questions about the child s behaviors and symptoms that might indicate such problems. Researchers want to see if the K-SADS-PL can help identify mental health problems in young adults (ages 18 to 25). Two groups of young adults, including healthy volunteers and people with cancer, and their parents will participate in this study.

Objectives:

* To see if the K-SADS-PL interview used for children and teens can also be used for young adults.
* To see whether information provided by parents will affect the rate of mental health problems found.

Eligibility:

* Individuals aged 18-25 years who have cancer and are participating in research studies at the National Institutes of Health.
* Healthy volunteers aged 18-25 years.
* A parent of a young adult who is participating in this study.

Design:

* This study requires one study visit that includes an interview and self-report questionnaires. It will take about 1 to 3 hours. A follow-up phone call or visit will also be required.
* Young adult participants will be given the K-SADS-PL interview and four questionnaires that ask about mood, anxiety, distress, parental contact, and development during childhood. The K-SADS-PL interview will be video recorded or audio recorded.
* Parents will also be given the K-SADS-PL interview. This interview can be done in person or by phone, and will also be recorded.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
Objective:

The goal of this pilot project is to describe the feasibility of using the Schedule for Affective Disorders and Schizophreni\a for School Age Children Present and Lifetime Version (K-SADS-PL) to screen and evaluate older adolescents and young adults (ages 18-25) for mood and anxiety disorders. An additional aim is to describe the contribution of the parent interview portion of the instrument for this age group. Two groups of 18-25 year old participants will be enrolled: healthy volunteers and patients with cancer. The information gained in this pilot study will inform the design of future intervention studies that target mood and anxiety disorders among pediatric oncology patients.

Primary aim:

Aim 1: Feasibility - Describe the feasibility of using the K-SADS-PL interview to screen and evaluate for mood and anxiety disorders among two groups of 18 25 year olds (healthy volunteers and patients with cancer) and their parents.

Hypothesis 1: The K-SADS-PL interview is feasible to use in the two groups of 18 25 year olds; the feasibility of completing the parent portion of the K-SADS-PL will be better among parents of cancer participants compared to parents of healthy volunteers.

Secondary aim:

Aim 2: K-SADS-PL outcomes - Compare and contrast K-SADS-PL findings based on responses provided by participants versus summary ratings that take into account both parent and child responses.

Hypothesis 2: Summary ratings of K-SADS-PL screening and diagnostic questions will yield more positive screening findings (subthreshold or threshold) compared to participant ratings alone.

Study population

This pilot study will include a convenience sample of young adults, aged 18-25, from two groups healthy volunteers and individuals who are participants in oncology protocols at the NIH Clinical Center (inpatient or outpatient) and who agree to participate. Participants may be from any institute, but must have a parent who will agree to be interviewed.

Design

This is a pilot study to describe the feasibility of extending the K-SADS-PL diagnostic interview to screen and evaluate young adults 18-25 years of age for psychiatric disorders. Informed consent will be obtained from the participant and his/her parent. The interview will be administered by a interviewer trained to administer the K-SADS-PL instrument. The same interviewer will administer the K-SADS-PLL to both the participant and the parent. The participant will be interviewed first, and the parent second. If there is more than one parent who is eligible, the parent who knows the participant best will be chosen. All interviews will be recorded. A subset of interview recordings will be randomly rated by a gold standard expert rater to determine inter-rater kappa coefficients for screening and diagnostic questions about mood and anxiety disorders.

Availability of parents to complete the K-SADS-PL interview will be optimized by allowing either face-to-face or phone interviews. If a parent interview reveals clinically significant information that the participant did not report, the interviewer will re-contact the participant to complete the necessary diagnostic module. Summary screening and diagnostic ratings will be determined by the interviewer, taking into account both participant and parent responses as per the K-SADS-PL design.

We will also ask participants to complete several short questionnaires:1) Hospital Anxiety and Depression Scale (HADS); 2) Parent-child frequency of contact; 3) Distress Thermometer; 4) Course of Life questionnaire.

ELIGIBILITY:
* a. Description of proband patients and healthy volunteers: these adult participants between the ages of 18-25 will be invited to undergo a psychiatric diagnostic interview using the K-SADS PL. Current or past history of mental health problems or treatment is allowed.

  b. Proband patient/healthy volunteer inclusion criteria
* Age 18-25 years, males and females
* English speaking
* Participant has contact (face-to-face, phone or electronic) with at least one of his/her parents at least once per week
* Enrolled in an NIH CC study (probands) or in good general health (healthy volunteers)

  c. Proband patient/healthy volunteer exclusion criteria
* Unable to provide informed consent
* Known severe intellectual disability such as a history of mental retardation, pervasive developmental disorder or inability to complete an 8th grade education.
* Initial cancer diagnosis within the past 3 months.
* Current unstable medical condition as evidenced by Karnofsky score below 50 (for cancer patients)
* Refusal to be video or audio recorded
* Cancer that involves the brain either as primary site of cancer or as a result of metastatic disease.

  d. Description of parent participants: If there is more than one parent who is eligible, the parent who knows the participant best will be chosen. For this study, we define parent as a primary caregiver during the participant s early life who directly observed the child s development and is still alive to be interviewed. This could allow for informants who are adoptive parents or other close relatives who raised the child.

  e. Parent participant inclusion criteria
* English speaking
* Parent of a patient proband or healthy volunteer enrolled in the study
* Parent has contact (face-to-face, phone or electronic) with his/her child at least once per week

  f. Parent participant exclusion criteria
* Unable to provide informed consent
* Known severe intellectual disability such as a history of mental retardation, pervasive developmental disorder or inability to complete an 8th grade education.
* Refusal to be video or audio recorded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01-26; Primary Completion 2016-08-25 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Feasibility defined in the 18-25 year old cancer patient group as a completion rate of greater than or equal to 60 percent among those approached to enter the study. | 2 years
Feasibility in parents is greater than or equal to 80 percent completion rate of the parent portion of the K-SADS-PL interview. | 2 years

SECONDARY OUTCOMES:
Frequency of positive (threshold or subthreshold) KSADS-PL summary ratings in both groups of participants. | 2 years
2x2 tables and kappa statistics that describe agreement between participant responses and summary ratings. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Y Chung, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ambrosini PJ. Historical development and present status of the schedule for affective disorders and schizophrenia for school-age children (K-SADS). J Am Acad Child Adolesc Psychiatry. 2000 Jan;39(1):49-58. doi: 10.1097/00004583-200001000-00016. PMID 10638067
- [Background] Birmaher B, Ehmann M, Axelson DA, Goldstein BI, Monk K, Kalas C, Kupfer D, Gill MK, Leibenluft E, Bridge J, Guyer A, Egger HL, Brent DA. Schedule for affective disorders and schizophrenia for school-age children (K-SADS-PL) for the assessment of preschool children--a preliminary psychometric study. J Psychiatr Res. 2009 Apr;43(7):680-6. doi: 10.1016/j.jpsychires.2008.10.003. Epub 2008 Nov 8. PMID 19000625
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252